CLINICAL TRIAL: NCT03353987
Title: Cognitive Training to Prevent Postoperative Cognitive Dysfunction in Older Patients - A Randomised Controlled Trial
Brief Title: Preoperative Cognitive Training for Postoperative Cognitive Dysfunction
Acronym: CogniTrain
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Patients are not compliant to the daily logbook exercises before surgery. Most will only perform once during training or maximum twice.
Sponsor: University of Malaya (Other)
Responsible Party: Principal Investigator, Dr Loh Pui San, Clinical Lecturer, University of Malaya
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2017312-5034
Record Dates: First submitted 2017-11-21; First posted 2017-11-27 (Actual); Last update posted 2019-08-05 (Actual); Status verified 2019-08

CONDITIONS: Cognitive Decline; Cognitive Impairment; Cognitive Deterioration
Keywords: Post-op cognitive dysfunction; Cognitive training; Logbook; Elderly
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Cognitive Training

STUDY DESIGN:
Intervention Model Description: Home based cognitive training (CogniTrain)
  Intervention: Using memory logbook and newspaper cuttings for cognitive improvement
Who Masked: Care Provider, Outcomes Assessor
Masking Description: The attending anaesthetist and assessors will be blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Preoperative counselling will be given upon recruitment Patients will be given instructions to continue their normal routine.
- Cognitive Training (Experimental): Preoperative counselling will be given upon recruitment Patients are taught cognitive training and are asked to perform a prescribed set of one-hour cognitive training daily for a minimum of 10 days and up to 1 month prior to surgery.
  Interventions: Behavioral: Cognitive training

INTERVENTIONS:
Behavioral: Cognitive training — Procedure
  1. A therapist will go through the daily routine of the participants at home before starting the intervention
  2. Selections of exercise items based on familiar items/ activities at home
  3. Given a memory logbook with list of household items, names and numbers and newspaper cuttings from the previous week
  4. Taught on how to perform the exercises
  5. Perform at least one hour per day
  6. Both spatial and visual memory strategies will be used for memory training: simple mnemonics, associations, visualisations, rhymes
  7. Advised to follow-up with the therapist to review on the progress and compliance of exercises weekly
  8. The difficulty of the exercise will be adjusted weekly
  List of exercises:
  1. Memorizing a set of lists, household items, names and numbers
  2. Summarising the contents of newspaper cuttings within a set of time
  3. Searching and listing sets of words from newspaper cuttings
  Other Names: Home based Cognive Training
  Arms: Cognitive Training

SUMMARY:
Postoperative Cognitive Dysfunction (POCD) is a state of decline in cognitive ability after surgery and is frequently seen among our elderly population. Many studies have looked into predictive risk factors for POCD while research is underway to search for pre-emptive measures to avoid this unfavourable outcome. Most will be looking at utilizing mobile software applications of cognitive training but in many poorer countries, owning electronic devices may not be an option or may be culturally less acceptable among the older patients. Hence, the investigators intend to investigate if a home-based logbook for cognitive training will reduce the incidence of POCD in a single centre study.

DETAILED DESCRIPTION:
Background:

Postoperative Cognitive Dysfunction (POCD) is a state in which a decline in cognitive ability after surgery persist from early postoperative period to a much longer term. It is said to be a subtle disorder of thought processes that influences domains of cognition such as memory especially short-term memory, inattention and inability to focus with the presence of generalized slowness. In fact, a lot of older patients and their loved ones claim they are 'never the same' after the surgery. It is to be distinguished from postoperative delirium, a diagnosis portrayed through several symptoms that occurs acutely after surgery, fluctuates with time and has a tendency to be transient. POCD, on the other hand, is difficult to diagnose and only detected by comparing postoperative results of neuropsychological battery tests to those done as baseline preoperatively.

Advanced age is a major risk for developing POCD.6 Studies done by the International Study of Postoperative Cognitive Dysfunction (ISPOCD) group had found an incidence of POCD at 19.2% within 1 week and 6.2% in 3 months. Similar studies have reported a higher figure of 36.1% at 1 week after surgery for this phenomenon. In certain high-risk groups, the range ascends to 16 - 62% with an average of 35% in hip fracture patients9 and up to 60% for those who underwent cardiac surgery that persist in 10-30% after 6 months.

Hypothesis:

As far as research is concerned, tremendous efforts are now underway to look for causes of POCD and its risk factors but most importantly, find ways to avoid this disability over time. Clinicians instinctively prescribe prehabilitation in preparation for surgery through various physical conditioning to improve patients' physiological cardio-respiratory reserve in the hope for better recovery. The investigators hypothesize that the same holds true with cognitive function and by optimizing mental 'fitness', the pre-conditioning can attribute to a decrease in POCD.

Currently, there are a few ongoing trials such as NeuroBics in US15 for non-cardiac surgery and Cog-train in UK for cardiac patients investigating the role of using electronic-based 'brain' intervention before surgery. The investigators aim to test the feasibility of using a home based logbook with easy applicability as the cognitive training to produce equally favourable results in reducing POCD since the socio-economic pattern of our older population is different from the west. Senior citizens may not be familiar with or have difficulty to afford electronic devices and are less engaged with web-based Internet as reflected by data from a local service provider that found only 3.9% of their user base in the country is over the age of 60.

Sample size:

Based on 36% POCD at one week from a previous study8 and our proposed 50% reduction to 18% incidence with intervention, a total of 232 participants (including 10% drop-out rate) are required at a 1:1 ratio between groups to achieve an 80% powered study and Type 1 error of 5%.

A preliminary analysis will be done at 50 recruited patients to look for feasibility of continuing this study.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 65 years of age or older, ASA I-III
2. Elective surgery (excluding neuro and cardiac surgery)
3. Date of surgery at least 10 days and up to one month from date of recruitment
4. Duration from induction of anaesthesia to end of anaesthesia minimum 2 hours
5. Expected post-operative hospital stay at least 48 hours
6. Able and willing to give informed consent
7. Literate
8. Willing to undergo cognitive and delirium assessments, perform daily cognitive training and able to return for follow-up assessments at 1 week, 3 months (phone call) and 1 year.

Exclusion Criteria:

1. Glasgow coma scale < 15
2. Geriatric depression score (GDS-5) ≥ 2
3. Pre-existing psychiatric disorder or delirium
4. Severe visual, hearing or speech impairment
5. General anaesthetic within the last 6 months

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 17 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2019-05-31 (Actual)

PRIMARY OUTCOMES:
Postoperative cognitive dysfunction | One week after surgery
  Any patient having deficit in 2 or more neuropsychological tests will be deemed to have POCD.
  A deficit in any test will be defined as a negative difference in scores and if the absolute value of each of these change scores is larger than one standard deviation (SD) of the baseline in the same cognitive test from all subjects. Any patient having deficit in 2 or more neuropsychological tests.
Postoperative cognitive dysfunction | One year after surgery
  Any patient having deficit in 2 or more neuropsychological tests will be deemed to have POCD.
  A deficit in any test will be defined as a negative difference in scores and if the absolute value of each of these change scores is larger than one standard deviation (SD) of the baseline in the same cognitive test from all subjects. Any patient having deficit in 2 or more neuropsychological tests.

SECONDARY OUTCOMES:
Identify age as a risk factor for developing POCD | One week and 1 year after surgery
  Correlation between patient age (in years) to POCD (Any patient having deficit in 2 or more neuropsychological tests will be deemed to have POCD.
  A deficit in any test will be defined as a negative difference in scores and if the absolute value of each of these change scores is larger than one standard deviation (SD) of the baseline in the same cognitive test from all subjects. Any patient having deficit in 2 or more neuropsychological tests.)
Identify the association between types of surgery performed with developing POCD | One week and 1 year after surgery
  Correlation between surgical procedures (orthopaedic/ general surgery/ ENT/ gynaecology) to POCD (Any patient having deficit in 2 or more neuropsychological tests will be deemed to have POCD.
  A deficit in any test will be defined as a negative difference in scores and if the absolute value of each of these change scores is larger than one standard deviation (SD) of the baseline in the same cognitive test from all subjects. Any patient having deficit in 2 or more neuropsychological tests.)
Identify the association between duration of anaesthesia with developing POCD | One week and 1 year after surgery
  Correlation between duration of anaesthesia (hours) to POCD (Any patient having deficit in 2 or more neuropsychological tests will be deemed to have POCD.
  A deficit in any test will be defined as a negative difference in scores and if the absolute value of each of these change scores is larger than one standard deviation (SD) of the baseline in the same cognitive test from all subjects. Any patient having deficit in 2 or more neuropsychological tests.)
Duration of home based cognitive training to prevent POCD | One week and 1 year after surgery
  Analysis of correlation between the total duration of cognitive training (hours) and incidence of POCD (Any patient having deficit in 2 or more neuropsychological tests will be deemed to have POCD.
  A deficit in any test will be defined as a negative difference in scores and if the absolute value of each of these change scores is larger than one standard deviation (SD) of the baseline in the same cognitive test from all subjects. Any patient having deficit in 2 or more neuropsychological tests.
Correlation between delirium and POCD | Post-op Day 1 to 3
  Analysis of correlation between positive CAM tests and incidence of POCD (Any patient having deficit in 2 or more neuropsychological tests will be deemed to have POCD.
  A deficit in any test will be defined as a negative difference in scores and if the absolute value of each of these change scores is larger than one standard deviation (SD) of the baseline in the same cognitive test from all subjects. Any patient having deficit in 2 or more neuropsychological tests.)

CONTACTS AND LOCATIONS:
Overall Officials: Pui San Loh, Principal Investigator — University of Malaya
Locations (1):
- University Malaya, Kuala Lumpur, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: Yes
Only IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Within 6 months after publication
Access Criteria: Written requests with supporting reasons to primary investigator for review among all investigators

REFERENCES:
- [Background] 1. Caza N. Progress in brain research 2008; 169: 409-22. 2. Deiner S. British journal of anaesthesia 2009; 103(suppl_1): i41-i6. 3. Wang W. Medical science monitor: international medical journal of experimental and clinical research 2014; 20: 1908. 4. Saniova B. Medical Science Monitor 2009; 15(5): CS81-CS7. 5. Cann C. Anaesthesia 2010; 65(12): 1166-9. 6. Monk TG. Anesthesiology: The Journal of the American Society of Anesthesiologists 2008; 108(1): 18-30. 7. Johnson T. The Journal of the American Society of Anesthesiologists 2002; 96(6): 1351-7. 8. Saleh AJ. Medical science monitor: international medical journal of experimental and clinical research 2015; 21: 798. 9. Bitsch M. Acta Orthopaedica Scandinavica 2004; 75(4): 378-89. 10. Newman MF. New England Journal of Medicine 2001; 344(6): 395-402. 11. Steinmetz J. Anaesthesia 2016; 71(S1): 58-63. 12. Hertzog C. Psychological science in the public interest 2008; 9(1): 1-65. 13. O'doherty A. British journal of anaesthesia 2013; 110(5): 679-89. 14. Kawano T. Anesthesiology: The Journal of the American Society of Anesthesiologists 2015; 123(1): 160-70. 15. Humeidan ML. . Clinical therapeutics 2015; 37(12): 2641-50.